CLINICAL TRIAL: NCT07400367
Title: Impact of a Multi-strain Probiotic Supplementation With Lifestyle Modification on Liver Steatosis, Fibrosis, and Metabolic Health in Patients With Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)
Brief Title: Impact of a Probiotic Supplementation With Lifestyle Modification on Liver Steatosis, Fibrosis, and Metabolic Health in Patients With Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FJUH114502
Record Dates: First submitted 2026-01-20; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Liver Elastography; Liver Steatosis; Liver Function Test; Insulin Resistance; Cardiometabolic Risk Factors
Keywords: MASLD; Probiotics; Liver fibrosis; Liver steatosis
MeSH Terms: conditions — Fatty Liver; Insulin Resistance; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receive the probiotic product one sachet per day and standard lifestyle modification education for MASLD by a gastroenterologist.
  Interventions: Dietary Supplement: Probiotic product; Behavioral: Life style modification
- Placebo (Active Comparator): Receive the placebo one sachet per day and standard lifestyle modification education for MASLD by a gastroenterologist.
  Interventions: Behavioral: Life style modification; Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Probiotic product — The probiotic product contains Lactobacillus salivarius AP-32, Lactobacillus rhamnosus bv-77, Bifidobacterium animalis CP-9 and Lactobacillus reuteri GL-104
  Arms: Intervention
Behavioral: Life style modification — Life style modification of MASLD provided by an gastroenterologist in an outpatient s
Dietary Supplement: placebo — placebo sachet looked and taste very similar to the probiotic product being tested
  Arms: Placebo

SUMMARY:
Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) is the new clinical term introduced in 2023 to redefine what was formerly known as Non-Alcoholic Fatty Liver Disease (NAFLD). It is defined as fatty liver confirmed by imaging or biopsy, accompanied by at least one cardiometabolic risk factor (e.g., hyperglycemia, dyslipidemia, hypertension, or obesity). Its pathological progression ranges from simple steatosis to steatohepatitis, primarily driven by excessive energy intake, hepatic lipid accumulation, and insulin resistance.

MASLD is currently the most prevalent chronic liver disease globally, with a prevalence rate of approximately 30-40%. However, there is no satisfactory pharmacological treatment, leaving lifestyle modification as the primary therapeutic approach. Many patients struggle to effectively adjust their habits, leading to persistent hepatic inflammation and damage, which may eventually progress to end-stage diseases such as cirrhosis and hepatocellular carcinoma. In many developed countries, MASLD has become the leading indication for liver transplantation, imposing a heavy burden on healthcare systems.

Gut dysbiosis is closely linked to MASLD. An imbalance in the gut microbiota disrupts the gut-liver axis, leading to impaired intestinal mucosal barrier function. This allows bacterial components to enter the circulation, further triggering hepatic inflammation and abnormal lipid metabolism. Consequently, modulating the gut microbiota is considered a potential therapeutic strategy.

Over the past decade, probiotics, prebiotics, and synbiotics have been extensively studied as non-pharmacological treatments for NAFLD. Multiple studies indicate that these products can reduce liver enzymes (AST, ALT), insulin resistance (HOMA-IR), and inflammatory markers (hs-CRP, TNF-α). The most effective combinations typically involve Lactobacillus, Bifidobacterium, and Streptococcus, with a recommended duration of approximately 12 weeks. However, the impact of these products on liver fibrosis, hepatic fat accumulation, and cardiometabolic risk factors remains inconclusive.

The probiotic product to be tested consists of Lactobacillus salivarius AP-32, Lactobacillus rhamnosus bv-77, Bifidobacterium animalis CP-9, and Lactobacillus reuteri GL-104. This formulation complies with food safety regulations. In clinical studies, it had been proven as an effective adjuvant method that increased beneficial gut bacteria such as Akkermansia muciniphila and improved the control of blood glucose, lipids, and inflammatory markers.

Study Objectives

This study aims to investigate the efficacy of this probiotic product as an adjuvant therapy alongside lifestyle modifications in adult patients with MASLD. We will evaluate its impact on:

1. The degree of liver fibrosis and steatosis
2. Cardiometabolic risk factors (BMI, waist circumference, blood lipids, and blood glucose).
3. Inflammatory markers.
4. Gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* ALT ≥ 60 U/L
* Liver steatosis identified by ultrasound
* Meet at least one cardiometabolic criteria:

  1. BMI ≥ 25 kg/m2 (Asian ≥23)
  2. Waist circumference: > 94cm (M) 80cm(F)
  3. Fasting blood glucose ≥ 100 mg/dL
  4. HbA1c ≥ 5.7
  5. Receiving treatment of diabetes
  6. Receiving treatment of Hypertension
  7. Average home blood pressure: ≥ 130/85 mmHg
  8. TG ≥ 150 mg/dL
  9. HDL ≤ 40 mg/dL
  10. Receiving treatment of dyslipidemia

Exclusion Criteria:

* HBsAg(+)
* Anti-HCV (+)
* Cirrhosis
* Excessive alcohol intake ( Male over 210g/wk; Female over 140mg/wk)
* Could not rule out Autoimmune hepatitis (ANA, or AMA or ASMA (+))
* Could not rule out drug related hepatitis
* Receiving drug that might induce liver steatosis:
* Glucocorticoids
* Amiodarone
* Tamoxifen
* Methotrexate
* Valproate
* Tetracycline
* Chemotherapeutic agents
* Receiving immune modulators or biologics
* Receiving antibiotics within 1 month
* Receiving any cancer treatment
* Have diagnosis of "Catastrophic Illness" defined by Health Administration of Taiwan
* eGFR<60
* Pregnancy
* Currently enrolled in other dietary or pharmacology clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in shear wave elastography (m/s) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in liver fibrosis at 12 weeks

SECONDARY OUTCOMES:
Change in ultrasound attenuation coefficient (dB/cm/MHz) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in liver steatosis at 12 weeks
Change in blood LDL level (mg/dL) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in blood LDL level (mg/dL) at 12 weeks
Change in blood HDL level (mg/dL) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in blood HDL level (mg/dL) at 12 weeks
Change in blood total cholesterol level (mg/dL) at 12 weeks | Time Frame: From enrollment to the end of treatment at 12 weeks
  Change in blood total cholesterol level (mg/dL) at 12 weeks
Change in blood triglycerides level (mg/dL) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in blood triglycerides level (mg/dL) at 12 weeks
Change in HOMA-IR at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in insulin resistance at 12 week
Change in blood fasting insulin level (μU/mL) at 12 weeks | From enrollment to the end of treatment at 12 weeks
Change in blood fasting glucose level (mg/dL) at 12 weeks | From enrollment to the end of treatment at 12 weeks
Change in blood AST level (U/L) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in liver function test
Change in blood ALT level (U/L) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in liver function test
Change in blood gamma-GT level (U/L) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in liver function tests
Change in blood alkaline phosphatase level (IU/L) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in liver function tests
Change in blood BUN level (mg/dL) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in renal function
Change in blood Creatinine level (mg/dL) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in renal functions
Change in eGFR level (mL/min/1.73m^2) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in renal function
Change in blood albumin level (g/dL) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in liver functions at 12 weeks
Change in platelet level (*10^3/uL) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  For the calculation of the chane of Fib-4 score at 12 weeks
Change in HbA1c level (%) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in blood sugar control at 12 weeks
Change in blood hs-CRP level (mg/L) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in systemic inflammation at 12 weeks
Change in blood IL-6 level (pg/mL) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in systemic inflammation at 12 weeks
Change in blood TNF-alpha level (pg/mL) at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in systemic inflammation at 12 weeks
Change in Fib-4 score at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in liver fibrosis score at 12 weeks
Change in ARPI score at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in liver fibrosis score at 12 weeks
Change in NAFLD Fibrosis Score at 12 weeks | From enrollment to the end of treatment at 12 weeks
  Change in liver fibrosis score at 12 weeks
Change in blood pressures (mmHg) at 12 weeks | From enrollment to the end of treatment at 12 weeks
Change in body weight (kg) at 12 weeks | From enrollment to the end of treatment at 12 weeks
Change in BMI (kg/m^2) at 12 weeks | From enrollment to the end of treatment at 12 weeks
Change in waist circumference (cm) at 12 weeks | From enrollment to the end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Jen Catholic University Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
de-identification data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Abhari K, Saadati S, Yari Z, Hosseini H, Hedayati M, Abhari S, Alavian SM, Hekmatdoost A. The effects of Bacillus coagulans supplementation in patients with non-alcoholic fatty liver disease: A randomized, placebo-controlled, clinical trial. Clin Nutr ESPEN. 2020 Oct;39:53-60. doi: 10.1016/j.clnesp.2020.06.020. Epub 2020 Jul 24. PMID 32859329
- [Background] Inoue K, Tsukuda S, Kayano H, Tanaka J, Heshiki A. A case of hypervascular renal capsule leiomyoma. Radiat Med. 2000 Sep-Oct;18(5):323-6. PMID 11128405
- [Background] Kumada T, Toyoda H, Ogawa S, Gotoh T, Yoshida Y, Yamahira M, Hirooka M, Koizumi Y, Hiasa Y, Tamai T, Kuromatsu R, Matsuzaki T, Suehiro T, Kamada Y, Sumida Y, Tanaka J, Shimizu M. Diagnostic performance of shear wave measurement in the detection of hepatic fibrosis: A multicenter prospective study. Hepatol Res. 2024 Sep;54(9):851-858. doi: 10.1111/hepr.14026. Epub 2024 Feb 13. PMID 38349813
- [Background] Farrow A, Farrow SC, Little R, Golding J. The repeatability of self-reported exposure after miscarriage. ALSPAC Study Team. Avon Longitudinal Study of Pregnancy and Childhood. Int J Epidemiol. 1996 Aug;25(4):797-806. doi: 10.1093/ije/25.4.797. PMID 8921459
- [Background] Jansson JH, Boman K, Brannstrom M, Nilsson TK. High concentration of thrombomodulin in plasma is associated with hemorrhage: a prospective study in patients receiving long-term anticoagulant treatment. Circulation. 1997 Nov 4;96(9):2938-43. doi: 10.1161/01.cir.96.9.2938. PMID 9386160
- [Background] Yang Y, Yang L, Wu J, Hu J, Wan M, Bie J, Li J, Pan D, Sun G, Yang C. Optimal probiotic combinations for treating nonalcoholic fatty liver disease: A systematic review and network meta-analysis. Clin Nutr. 2024 Jun;43(6):1224-1239. doi: 10.1016/j.clnu.2024.04.004. Epub 2024 Apr 13. PMID 38643738
- [Background] Wu J, Chen X, Qian J, Li G. Clinical improvement effect of regulating gut microbiota on metabolic dysfunction-associated steatotic liver disease: Systematic review and meta-analysis of randomized controlled trials. Clin Res Hepatol Gastroenterol. 2024 Aug;48(7):102397. doi: 10.1016/j.clinre.2024.102397. Epub 2024 Jun 13. PMID 38879003
- [Background] Sharma S, Tiwari N, Tanwar SS. The current findings on the gut-liver axis and the molecular basis of NAFLD/NASH associated with gut microbiome dysbiosis. Naunyn Schmiedebergs Arch Pharmacol. 2025 Sep;398(9):11541-11579. doi: 10.1007/s00210-025-04069-z. Epub 2025 Apr 9. PMID 40202676
- [Background] Ledru E, Diagbouga S, Tranchot-Diallo J, Cauchoix B, Yameogo M, Chami D, Soula G, Chiron JP. Eosinophils: a putative marker of immunodepression in HIV-infected African patients with tuberculosis? Trans R Soc Trop Med Hyg. 1994 Jan-Feb;88(1):117-8. doi: 10.1016/0035-9203(94)90531-2. No abstract available. PMID 7908766
- [Background] Su X, Chen S, Liu J, Feng Y, Han E, Hao X, Liao M, Cai J, Zhang S, Niu J, He S, Huang S, Lo K, Zeng F. Composition of gut microbiota and non-alcoholic fatty liver disease: A systematic review and meta-analysis. Obes Rev. 2024 Jan;25(1):e13646. doi: 10.1111/obr.13646. Epub 2023 Oct 9. PMID 37813400